CLINICAL TRIAL: NCT01109797
Title: A Comparison of Two Models for Transition of Adolescents and Young Adults With Diabetes From Pediatric to Adult Care
Brief Title: Transition of Adolescents and Young Adults With Diabetes From Pediatric to Adult Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12157
Record Dates: First submitted 2010-04-19; First posted 2010-04-23 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transition Social Behavioral Intervention (Experimental)
  Interventions: Behavioral: Transition Social Behavioral Intervention
- Diabetes Transition Clinic (Experimental)
  Interventions: Behavioral: Diabetes Transition Clinic

INTERVENTIONS:
Behavioral: Transition Social Behavioral Intervention — If you are assigned to the first group, you will have two all-day Saturday sessions four weeks apart on the KU campus in Lawrence. The objectives of the Saturday programs are to promote positive behavior change with respect to "taking ownership" of diabetes and its demands by providing transition-specific information, enabling participants to practice the life skills needed to successfully manage diabetes as an adult, and fostering peer-to-peer social networking over the 6-month period of the intervention (and beyond). You will continue to see your current provider of diabetes care outside of the parameters of this study.
  Arms: Transition Social Behavioral Intervention
Behavioral: Diabetes Transition Clinic — Patients who participate in the transition clinic arm of the study will be seen six times during a six-month time period, as well as receive psychological assessment and intervention, as necessary, prior to the first clinic visit (intake) and as part of visits 2 and 4. Three of the six visits will be standard of care medical visits with either a pediatric or adult provider or both. Three will be individual or group education sessions with diabetes educators focused on transition issues such as, managing the adult health care system, talking with your care provider,and dealing with adult issues (pregnancy, genetic concerns, etc).
  Arms: Diabetes Transition Clinic

SUMMARY:
The purpose of the study is to compare two interventions for preparing diabetic teens and young adults for transition from pediatric to adult diabetes care.

DETAILED DESCRIPTION:
One will represent a short-term intensive social-behavioral intervention supported by peer-to-peer social networking in which subjects receive "usual care" from their current diabetes provider outside the parameters of the study. The second intervention will be a traditional transition clinic model, where subjects will receive the standard of diabetes care from a team of combined pediatric and adult practitioners and educators, with added educational modules and behavioral evaluation and support designed to facilitate the transition to adult care (i.e., that foster "developmentally tailored care"). The first is a much less intensive intervention from the standpoint of the providers and gives special prominence to peer support; the second is provider-intensive. The goal of both interventions is to improve self-efficacy (confidence in taking ownership of and managing one's diabetes); i.e., to prepare the patient to move from primary support by family and providers to a reliance on self-ownership and self-management as a responsible, independent adult.

Optional sub-study available for parents, spouses, and significant others.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-29
* Diagnosis of type 1 diabetes, or type 2 diabetes managed with insulin, at least one year prior to study initiation
* English-speaking
* Some form of private or public (e.g., Medicaid) health insurance

Exclusion Criteria:

* Cystic fibrosis-related or pancreatitis-related diabetes
* Diabetes related to a known specific genetic defect such as Down's Syndrome, Lipoatrophic Diabetes, Leprechaunism or Rabson-Mendenhall Syndrome, etc.
* Chronic liver disease
* History of chronic renal failure
* Serious psychiatric illness that in the judgment of the investigators would preclude the individual's ability to complete the study
* Pregnant or planning to become pregnant within 6 months

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Measure and compare change in self-efficacy and change in diabetes knowledge, diabetes quality of life, family conflict, and treatment satisfaction for and between the two groups. | 6 months and 12 months

SECONDARY OUTCOMES:
Make exploratory baseline comparisons between the two groups regarding locus of diabetes care (kind of provider), comparing numbers of subjects in each group who made a successful transition to adult care | 6 months and 12 months
Make exploratory baseline comparisons between the two groups of using some form of social networking by the two groups as an adjunt of diabetes care. | 6 months and 12 months
Make exploratory baseline comparisons between the two groups regarding provider and educator time devoted in each arm of the intervention (in order to prepare for a robust comparative effectiveness analysis in a subsequent study). | 6 months
Make exploratory baseline comparisons between the two groups of HgbA1c | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Midyett, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States